CLINICAL TRIAL: NCT01904487
Title: Characterization of [11C]Flumazenil to Image GABA Transmission in Healthy Adult Subjects and Subjects With Alcohol Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rajesh Narendran (Other)
Responsible Party: Sponsor-Investigator, Rajesh Narendran, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO#10100519
Record Dates: First submitted 2013-07-16; First posted 2013-07-22 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Tiagabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET scans (Experimental): Both alcoholics and healthy controls will undergo two [11C]flumazenil PET scans: one at baseline and one post administration of 0.2 mg/kg Tiagabine.
  Interventions: Radiation: [11C]flumazenil; Drug: Tiagabine

INTERVENTIONS:
Radiation: [11C]flumazenil — [11C]flumazenil is a radiotracer used to measure levels of the neurotransmitter GABA in the human brain.
Drug: Tiagabine — Tiagabine raises levels of GABA in the brain. It is used in this study so that we can measure the changes in GABA levels.

SUMMARY:
Background:

- This study is being done to examine the role of a chemical GABA in the brain of alcohol dependent patients. GABA is the chief inhibitory neurotransmitter in the central nervous system. It helps induce relaxation and sleep and balances the brain by inhibiting over-excitation. Several studies have reported that anxiety disorders such as panic attacks, seizure disorders, and numerous other conditions including addiction, are all related to low GABA activity. Therefore, we will examine differences in GABA levels between healthy controls and subjects with alcohol addiction. Studies such as this are important to the understanding of the role of GABA in alcohol addiction.

DETAILED DESCRIPTION:
Objectives:

- By comparing the two PET scans (before and after tiagabine) done in the same day, we can understand more about how much GABA your brain makes and about the activity of your GABA receptors in the brain.

Eligibility:

- Individuals 18-45 years of age who are heavy drinkers or healthy controls.

Design:

* Procedures to determine if you are eligible to take part in a research study are called "screening procedures". This will require you to come to the investigators office for approximately ½ day. For this research study, the screening procedures include comprehensive psychiatric and medical evaluations. Participants be asked to abstain from drugs and alcohol for the duration of the study and will be required to make trips several times a week for two weeks to provide clean urine samples.
* During one of the visits prior to the PET scans, participants will have a magnetic resonance image (MRI) taken of their brain.
* We will be using a technology called Positron Emission Tomography (PET), which is a method used to take pictures of the body, in this case, the brain. We will be injecting you with a radiotracer called [11C]flumazenil. A radiotracer is a small amount of a drug with radioactivity attached. Because the radiotracer temporarily sticks to the GABA receptors in the brain, the PET scan can then measure the activity at GABA receptors by measuring the amount of the radiotracer. You will undergo two PET scans with [11C]flumazenil on one day for this study. After the first PET scan, you will be given an oral dose of tiagabine (Gabitril®), which is a medication approved for the treatment of seizure disorder. Tiagabine raises levels of GABA in the brain. It is used in this study so that we can measure the changes in GABA levels. Blood samples will be drawn during the PET scans.

ELIGIBILITY:
Inclusion Criteria:

Healthy Control Subjects:

1. Males or Females 18-45
2. Absence of present or past psychiatric conditions (including alcohol or drug dependence)
3. A negative urine drug screen
4. Medically Healthy

Subjects with alcohol dependence:

1. Males or Females 18-45
2. Fulfill DSM-IV Diagnosis for Alcohol Dependence
3. Negative Urine Drug Screen
4. Negative Urine ETG/ETS
5. Medically Healthy
6. Abstinent from alcohol for a minimum of 1 month prior to scanning procedures

Exclusion Criteria:

Healthy Control Subjects:

1. Pregnancy or lactation, lack of effective birth control during 15 days before the scans
2. Presence or positive history of serious medical or neurological illness, including low hemoglobin.
3. Any use (within recent past 6 weeks) of amphetamines, opiates, cocaine, ecstasy PCP.
4. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan (but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant. Dental fillings do not present a risk for MRI), as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists.
5. Currently employed as radiation worker; or participation in radioactive drug research protocols within the previous year such that the total cumulative annual radiation dose (i.e., from participation in the previous research studies and this study) would exceed the radiation dose limits specified in the FDA regulations at 21 CFR 361.1, Radioactive Drugs Considered Generally Safe and Effective (i.e. annual cumulative radiation dose limit = 5 rems to gonads, blood-forming organs, lens of eye, whole body; 15 rems to other organs).
6. Subjects with known hypersensitivity to flumazenil or benzodiazepines; subjects who have been given a benzodiazepine for control of a potentially life-threatening condition (e.g., control of intracranial pressure or status epilepticus or in patient who are showing signs of serious cyclic antidepressant overdose)

Subjects with alcohol dependence:

1. Pregnancy or lactation, lack of effective birth control during 15 days before the scans
2. Presence or positive history of serious medical or neurological illness or any cardiovascular disease, low hemoglobin
3. Any other current major axis I psychiatric diagnosis except alcohol dependence (subjects with nicotine dependence will not be excluded)
4. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan (but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant. Dental fillings do not present a risk for MRI), as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists.
5. Currently employed as radiation worker; or participation in radioactive drug research protocols within the previous year such that the total cumulative annual radiation dose (i.e., from participation in the previous research studies and this study) would exceed the radiation dose limits specified in the FDA regulations at 21 CFR 361.1, Radioactive Drugs Considered Generally Safe and Effective (i.e. annual cumulative radiation dose limit = 5 rems to gonads, blood-forming organs, lens of eye, whole body; 15 rems to other organs).
6. Subjects with known hypersensitivity to flumazenil or benzodiazepines; subjects who have been given a benzodiazepine for control of a potentially life-threatening condition (e.g., control of intracranial pressure or status epilepticus or in patient who are showing signs of serious cyclic antidepressant overdose)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-04-19; Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-01 (Actual)

PRIMARY OUTCOMES:
To measure changes in [11C]flumazenil binding in the brain using PET scans | Day 1: baseline PET scan and a follow-up PET scan 0.5 hours post administration of Tiagabine
Tiagabine induced change in [C-11]flumazenil distribution volume (VT) | 1 hour
  Refer to for consensus nomenclature J Cereb Blood Flow Metab. 2007 Sep;27(9):1533-9. Epub 2007 May 9.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Narendran, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Lingford-Hughes AR, Wilson SJ, Cunningham VJ, Feeney A, Stevenson B, Brooks DJ, Nutt DJ. GABA-benzodiazepine receptor function in alcohol dependence: a combined 11C-flumazenil PET and pharmacodynamic study. Psychopharmacology (Berl). 2005 Aug;180(4):595-606. doi: 10.1007/s00213-005-2271-x. Epub 2005 Apr 28. PMID 15864554
- [Background] Gilman S, Adams KM, Johnson-Greene D, Koeppe RA, Junck L, Kluin KJ, Martorello S, Heumann M, Hill E. Effects of disulfiram on positron emission tomography and neuropsychological studies in severe chronic alcoholism. Alcohol Clin Exp Res. 1996 Nov;20(8):1456-61. doi: 10.1111/j.1530-0277.1996.tb01149.x. PMID 8947325
- [Background] Farde L, Pauli S, Litton JE, Halldin C, Neiman J, Sedvall G. PET-determination of benzodiazepine receptor binding in studies on alcoholism. EXS. 1994;71:143-53. doi: 10.1007/978-3-0348-7330-7_15. PMID 8032146
- [Background] Litton JE, Neiman J, Pauli S, Farde L, Hindmarsh T, Halldin C, Sedvall G. PET analysis of [11C]flumazenil binding to benzodiazepine receptors in chronic alcohol-dependent men and healthy controls. Psychiatry Res. 1993 Apr;50(1):1-13. doi: 10.1016/0925-4927(93)90019-e. PMID 8390063
- See also: Psychiatric Molecular Imaging Program Addiction Website — http://www.addictionstudies.pitt.edu/